CLINICAL TRIAL: NCT00718588
Title: A Phase I, Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial, With a Single Ascending-Dose Stage Followed by a Multiple Ascending-Dose Stage, of the Safety, Pharmacokinetics, and Pharmacodynamics of Intravenous and Subcutaneous MTRX1011A in Patients With Rheumatoid Arthritis
Brief Title: A Study of the Safety, Pharmacokinetics, and Pharmacodynamics of MTRX1011A in Patients With Rheumatoid Arthritis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study had completed enrollment but drug injection was halted due to an unacceptable incidence of rash.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDT4478g
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Rheumatoid Arthritis
Keywords: RA
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MTRX1011A — Subcutaneous and intravenous single and repeating dose

SUMMARY:
This is a Phase I multicenter study that will be conducted in the United States and consists of a double-blind, placebo-controlled, SAD stage, followed by a double-blind, placebo controlled MAD stage. The study will be conducted in approximately 65 adult patients between 18 and 80 years old who have RA.

ELIGIBILITY:
Inclusion Criteria:

1. SAD Stage

   * RA diagnosed according to the ACR
   * For patients taking anti-rheumatic therapies, receipt of a stable regimen prior to randomization
   * Previous treatment with biologic agents, including anti-TNF agents, permitted but discontinued for an appropriate washout period
2. MAD Stage (same as above with the addition of the following)

   * Failure of at least one biologic agent, defined as lack of or loss of response or intolerance
   * Active disease defined by swollen and tender count

Exclusion Criteria:

* Significant systemic involvement of RA, including vasculitis, pulmonary fibrosis, or Felty's syndrome
* Malignancy, or prior malignancy, other than non-melanoma skin cancer or cervical carcinoma in situ that has been resected
* History of treatment with any T cell-directed therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-07; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of MTRX1011A in both the SAD and MAD stages | Length of study

SECONDARY OUTCOMES:
Characterize the pharmacokinetic response of MTRX1011A | Length of study
Characterize the pharmacodynamic profile of single and multiple doses of MTRX1011A | Length of study

CONTACTS AND LOCATIONS:
Overall Officials: John Davis, M.D., M.P.H., Study Director — Genentech, Inc.